CLINICAL TRIAL: NCT00146536
Title: The Incidence of Adjacent Synchronous Ipsilateral Infiltrating Carcinoma, DCIS, or Atypical Ductal Hyperplasia (ADH) in Patients Diagnosed With Lobular Neoplasia of the Breast by Core Needle Biopsy
Brief Title: Upstaging of ALH/LCIS Found on Core Biopsy Based on Subsequent Excisional Biopsy
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Faina Nakhlis, MD, Instructor in Surgery, Harvard Medical School, Dana-Farber Cancer Institute
Other Study IDs: 04-164
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2012-11

CONDITIONS: Breast Neoplasms
Keywords: ALH; LCIS; DCIS; adjacent ipsilateral infiltrating carcinoma; core needle biopsy; Lobular neoplasia of the breast
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Option of keeping tissue sample for further research
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to determine how often patients who have atypical lobular hyperplasia (ALH) or lobular carcinoma in situ (LCIS) on core needle biopsy of an imaging (found by mammogram or breast ultrasound) abnormality will have associated breast cancer at surgical removal of the area.

DETAILED DESCRIPTION:
Patients will undergo a breast biopsy at which the area found to be ALH or LCIS on core biopsy will be removed surgically through a small incision in the breast.

* The surgical biopsy specimen will be carefully examined by a pathologist, and may be useful in guiding further therapy if needed.
* In the future, tissue from the surgical biopsy may be used to study genetic changes that may be responsible for cancer formation and prevention. The tissue will be kept for future research for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Women 20 years of age or older
* Imaging abnormality necessitating a core needle biopsy
* Core needle biopsy revealing ALH or LCIS
* Patients may have a history of fibroadenoma and/or proliferative breast lesions with atypia

Exclusion Criteria:

* History and/or concomitant diagnosis of invasive breast cancer or ductal carcinoma in situ (DCIS)
* A palpable abnormality diagnosed by core needle biopsy to be ALH or LCIS
* Received tamoxifen in the past

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have ALH/LCIS detected on a needle biospy of the breast
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2004-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Rate of upstaging from Lobular Neoplasia on core biopsy to invasive breast cancer or ductal carcinoma in situ on excisional biopsy | Concomittant

SECONDARY OUTCOMES:
Factors which predict for upstaging from Lobular Neoplasia on core biopsy to invasive breast carcinoma or ductal carcinoma in situ

CONTACTS AND LOCATIONS:
Overall Officials: Faina Nakhlis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts